CLINICAL TRIAL: NCT03273920
Title: Robotic Versus Laparoscopic Distal Gastrectomy With D2 Lymphadenectomy for Locally Advanced Gastric Cancer: a Multicenter Randomized Controlled Trial
Brief Title: Robotic Versus Laparoscopic Distal Gastrectomy With D2 Lymphadenectomy for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Collaborators: Chinese PLA General Hospital (Other); West China Hospital (Other); Xijing Hospital of Digestive Diseases (Other); Nanjing PLA General Hospital (Other); Peking University Cancer Hospital & Institute (Other); Qingdao University (Other); Fujian Medical University Union Hospital (Other); Central South University (Other); The First Affiliated Hospital of Nanchang University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Jilin Provincial Tumor Hospital (Other); Lanzhou General Hospital of PLA (Other)
Responsible Party: Principal Investigator, Yan Shi, Deputy director, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRASS-01
Record Dates: First submitted 2017-08-23; First posted 2017-09-06 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Gastric Cancer
Keywords: laparoscopy-assisted gastrectomy; robot-assisted gastrectomy; advanced gastric cancer; D2 Lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic gastrectomy (Experimental): Robotic distal gastrectomy with D2 nodal dissection
  Interventions: Procedure: Robotic distal gastrectomy with D2 nodal dissection
- Laparoscopic gastrectomy (Active Comparator): Laparoscopic distal gastrectomy with D2 nodal dissection
  Interventions: Procedure: Laparoscopic distal gastrectomy with D2 nodal dissection

INTERVENTIONS:
Procedure: Robotic distal gastrectomy with D2 nodal dissection — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, robotic distal gastrectomy with D2 lymph node dissection will be performed with curative treated intent.The type of reconstruction will be determined by the surgeon's experience and preference. The reconstruction can be carried out by extracorporeal or intracorporeal anastomosis.
  Arms: Robotic gastrectomy
Procedure: Laparoscopic distal gastrectomy with D2 nodal dissection — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, laparoscopic distal gastrectomy with D2 lymph node dissection will be performed with curative treated intent.The type of reconstruction will be determined by the surgeon's experience and preference. The reconstruction can be carried out by extracorporeal or intracorporeal anastomosis.
  Arms: Laparoscopic gastrectomy

SUMMARY:
This study is an investigator-initiated, randomized, controlled, parallel group, and non-inferiority trial comparing robot-assisted gastrectomy with D2 nodal dissection for locally advanced gastric cancer patients with laparoscopic procedure.

DETAILED DESCRIPTION:
Since the first case of laparoscopy-assisted distal gastrectomy was reported in 1994, the number of patients undergoing the laparoscopic procedure has gradually increased. The latest Japanese gastric cancer treatment guideline recommends laparoscopic gastrectomy (LG) as an optional treatment for cStage I gastric cancer (GC). Based on the experience of early GC, most experienced surgeons have applied the laparoscopic procedure in patients with locally advanced gastric cancer (AGC). According to the results of large-scaled retrospective studies and ongoing randomized controlled trials (RCTs), LG treating AGC can gain better short-term outcomes and comparable long-term oncologic results.

To minimize the limitations of laparoscopic surgery, robot systems have been introduced to treat GC providing technical advantages. Though the feasibility and safety of robotic gastrectomy (RG) have been well accepted, the benefits of RG remain controversial. A recent meta-analysis including eleven studies of 3503 patients demonstrated that RG indicated potentially favorable outcomes in terms of blood loss compared with LG. Furthermore, it has been confirmed that robotic system could provide an advantage over LG in the dissection of the N2 area lymph nodes, especially around the splenic artery area. Our previous study demonstrated that the RG had less intraoperative blood loss and more lymph nodes dissection compared with the laparoscopic procedure. However, the only prospective study reported that RG is not superior to LG in terms of perioperative surgical outcomes. Nevertheless, the following subgroup analysis found that patients with GC undergoing D2 lymph node dissection can benefit from less blood loss when a robotic surgery system is used. Take together, RG with D2 nodal dissection may be superior laparoscopic surgery in terms of blood loss and retrieved lymph nodes. However, lack of high-level evidence-based medical researches, we can't drew a conclusion that patients with AGC may benefit from RG with D2 nodal dissection.

With regard to a new surgical approach, oncologic safety has attracted more attention. Although some retrospective studies have demonstrated that RG with lymphadenectomy for GC had non-inferior oncologic outcome relative to LG, there is no prospective RCT to evaluate the long-term outcomes of RG. Therefore, the Chinese Robotic Gastrointestinal Surgery Study (CRASS) Group launched a multicenter prospective RCT to verify the short-term and long-term outcomes of RG in AGC. The primary objective of this study is to assess whether robot-assisted distal gastrectomy is comparable to laparoscopic approach in terms of long-term oncologic outcomes without compromising relapse-free survival. The secondary research objectives are to compare robotic and laparoscopic approach in terms of morbidity, mortality, quality of life, cost-effectiveness, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven gastric adenocarcinoma.
2. Tumor located in the lower third of the stomach, and is possible to be curatively resected by subtotal gastrectomy.
3. Preoperative stage of cT2-4aN0-3M0 according to American Joint Committee on Cancer/Union for International Cancer Control 8th edition
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. American Society of Anesthesiology (ASA) score of class I to III
6. Patients who freely give informed consent to participate in the clinical study

Exclusion Criteria:

1. Previous upper abdominal surgery (except laparoscopic cholecystectomy)
2. Previous gastric resection (gastrectomy, endoscopic mucosal resection, or endoscopic submucosal dissection)
3. Gastric cancer-related complications (complete obstruction or perforation)
4. Enlarged or bulky regional lymph node diameter larger than 3 cm based on preoperative imaging
5. Previous neoadjuvant chemotherapy or radiotherapy for gastric cancer
6. Patients diagnosed with other malignancy within 5 years
7. Severe mental disorder
8. Unstable angina or myocardial infarction within the past 6 months
9. Cerebrovascular accident within the past 6 months
10. Severe respiratory disease (FEV1< 50%)
11. Continuous systemic steroid therapy within 1 month before the study
12. Pregnant or breast-feeding women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1110 (Estimated)
Dates: Start 2017-09-25 (Estimated); Primary Completion 2019-09-25 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
3-year relapse-free survival | 3 years
  Relapse-free survival is defined as days from surgery to recurrence or death from any cause, and it is censored at the latest day when the patient is alive without any evidence of recurrence.

SECONDARY OUTCOMES:
Morbidity | 30 days
  Early postoperative morbidity confined to events that occur within 30 days after surgery. The complications that occur after postoperative day 30 belong to late postoperative morbidity
Mortality | 30 days
  Postoperative mortality is defined to death that occurs within 30 days.
3-year overall survival | 3 years
  Overall survival is defined as days from surgery to death from any cause, and it is censored at the last day when the patient was alive.
3-year recurrence pattern | 3 years
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Postoperative recovery course | 15 days
  Time to first ambulation, flatus, liquid diet, soft diet, and duration of hospital stay are used to assess the postoperative recovery course.
Inflammatory response | 7 days
  The daily highest body temperature before discharge and the values of white blood cell count (10^9/L), hemoglobin (g/L), C-reactive protein (mg/L) and prealbumin (mg/L) from peripheral blood before operation and on postoperative day 1, 3, 5, 7 are recorded.
Immune response | 7 days
  The values of relevant immune cytokines from peripheral blood before operation and on postoperative day 1, 3, 5, 7 are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Peiwu Yu, M.D., Study Chair — Southwest Hospital, China
Locations (14):
- China (14):
  - Chinese PLA general hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Department of General Surgery and Center of Microinvasive Gastrointestinal Surgery, Southwest Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Lanzhou PLA General Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing General Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Xijing Hospital of Digestive Dieases, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Zhao Y, Yu P, Hao Y, Qian F, Tang B, Shi Y, Luo H, Zhang Y. Comparison of outcomes for laparoscopically assisted and open radical distal gastrectomy with lymphadenectomy for advanced gastric cancer. Surg Endosc. 2011 Sep;25(9):2960-6. doi: 10.1007/s00464-011-1652-y. Epub 2011 Apr 22. PMID 21512884
- [Background] Hu Y, Ying M, Huang C, Wei H, Jiang Z, Peng X, Hu J, Du X, Wang B, Lin F, Xu J, Dong G, Mou T, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Oncologic outcomes of laparoscopy-assisted gastrectomy for advanced gastric cancer: a large-scale multicenter retrospective cohort study from China. Surg Endosc. 2014 Jul;28(7):2048-56. doi: 10.1007/s00464-014-3426-9. Epub 2014 Mar 21. PMID 24651893
- [Background] Hu Y, Huang C, Sun Y, Su X, Cao H, Hu J, Xue Y, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Chen P, Liu H, Zheng C, Liu F, Yu J, Li Z, Zhao G, Chen X, Wang K, Li P, Xing J, Li G. Morbidity and Mortality of Laparoscopic Versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Apr 20;34(12):1350-7. doi: 10.1200/JCO.2015.63.7215. Epub 2016 Feb 22. PMID 26903580
- [Background] Inaki N, Etoh T, Ohyama T, Uchiyama K, Katada N, Koeda K, Yoshida K, Takagane A, Kojima K, Sakuramoto S, Shiraishi N, Kitano S. A Multi-institutional, Prospective, Phase II Feasibility Study of Laparoscopy-Assisted Distal Gastrectomy with D2 Lymph Node Dissection for Locally Advanced Gastric Cancer (JLSSG0901). World J Surg. 2015 Nov;39(11):2734-41. doi: 10.1007/s00268-015-3160-z. PMID 26170158
- [Background] Hashizume M, Shimada M, Tomikawa M, Ikeda Y, Takahashi I, Abe R, Koga F, Gotoh N, Konishi K, Maehara S, Sugimachi K. Early experiences of endoscopic procedures in general surgery assisted by a computer-enhanced surgical system. Surg Endosc. 2002 Aug;16(8):1187-91. doi: 10.1007/s004640080154. Epub 2002 May 3. PMID 11984681
- [Background] Junfeng Z, Yan S, Bo T, Yingxue H, Dongzhu Z, Yongliang Z, Feng Q, Peiwu Y. Robotic gastrectomy versus laparoscopic gastrectomy for gastric cancer: comparison of surgical performance and short-term outcomes. Surg Endosc. 2014 Jun;28(6):1779-87. doi: 10.1007/s00464-013-3385-6. Epub 2014 Jan 3. PMID 24385251
- [Background] Nakauchi M, Suda K, Susumu S, Kadoya S, Inaba K, Ishida Y, Uyama I. Comparison of the long-term outcomes of robotic radical gastrectomy for gastric cancer and conventional laparoscopic approach: a single institutional retrospective cohort study. Surg Endosc. 2016 Dec;30(12):5444-5452. doi: 10.1007/s00464-016-4904-z. Epub 2016 Apr 29. PMID 27129542
- [Background] Obama K, Kim YM, Kang DR, Son T, Kim HI, Noh SH, Hyung WJ. Long-term oncologic outcomes of robotic gastrectomy for gastric cancer compared with laparoscopic gastrectomy. Gastric Cancer. 2018 Mar;21(2):285-295. doi: 10.1007/s10120-017-0740-7. Epub 2017 Jun 21. PMID 28639136
- [Background] Duan BS, Zhao J, Xie LF, Wang Y. Robotic Verse Laparoscopic Gastrectomy for Gastric Cancer: A Pooled Analysis of 11 Individual Studies. Surg Laparosc Endosc Percutan Tech. 2017 Jun;27(3):147-153. doi: 10.1097/SLE.0000000000000410. PMID 28582378
- [Background] Kim HI, Han SU, Yang HK, Kim YW, Lee HJ, Ryu KW, Park JM, An JY, Kim MC, Park S, Song KY, Oh SJ, Kong SH, Suh BJ, Yang DH, Ha TK, Kim YN, Hyung WJ. Multicenter Prospective Comparative Study of Robotic Versus Laparoscopic Gastrectomy for Gastric Adenocarcinoma. Ann Surg. 2016 Jan;263(1):103-9. doi: 10.1097/SLA.0000000000001249. PMID 26020107
- [Background] Park JM, Kim HI, Han SU, Yang HK, Kim YW, Lee HJ, An JY, Kim MC, Park S, Song KY, Oh SJ, Kong SH, Suh BJ, Yang DH, Ha TK, Hyung WJ, Ryu KW. Who may benefit from robotic gastrectomy?: A subgroup analysis of multicenter prospective comparative study data on robotic versus laparoscopic gastrectomy. Eur J Surg Oncol. 2016 Dec;42(12):1944-1949. doi: 10.1016/j.ejso.2016.07.012. Epub 2016 Jul 29. PMID 27514719